CLINICAL TRIAL: NCT06143137
Title: Recovery From Acute Immune Failure in Septic Shock by Immune Cell Extracorporeal Therapy - Observational Long-term Outcome Follow up
Acronym: ReActIF- LTO
Status: Recruiting | Type: Observational
Sponsor: Artcline GmbH (Industry)
Collaborators: ZKS Jena (Unknown)
Responsible Party: Sponsor
Other Study IDs: ReActIF-ICE-LTO_ZKSJ0154
Record Dates: First submitted 2023-08-08; First posted 2023-11-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2023-08

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Subjects in this group where randomized in the control group in the ReActiF-ICE study previously
- Therapy Group: Subjects in this group where randomized in the therapy group in the ReActiF-ICE study previously

SUMMARY:
Subjects previously enrolled / randomized in the ReActIF-ICE (Recovery from acute immune failure in septic shock by immune cell extracorporeal terapy - immune competence enhancement) study received either standard sepsis treatment (control group) or standard sepsis treatment and additionally the ARTICE treatment (treatment group) during their index hospitalization. All subjects are followed up for 90 days after enrollment.

In this long term follow up study, the enrolled subjects shall be followed up beyond 90 days for up to 5 years.

DETAILED DESCRIPTION:
Sepsis is a worldwide health threat because of high mortality and the development of long-lasting disabilities, including physical and cognitive impairment and mental disorders, known collectively as post-intensive care syndrome (PICS), which contribute to reduced health-related quality of life (HRQoL) for several years even after successful recovery from the initial acute sepsis state. Sepsis survivors often need a longer period of rehabilitation, consuming more medical and social resources and struggle with financial burdens.

In the ReActIF-ICE study, that started enrolling patients in July 2022, up to 142 subjects with severe sepsis are to be enrolled and randomized into a therapy group (receiving the ARTICE treatment (extracorporeal immune cell plasma perfusion) on top of standard care) and control group (standard care only). These subjects were followed up according the ReActIF-ICE study protocol for 90 days.

Since there is still a large need for long-term outcome data of sepsis patients, collecting data of the ReActIF-ICE patients over a longer period of time would provide important additional information regarding:

1. General long term clinical and socio-economic outcome of sepsis survivors
2. Long-term outcome details of the ReActIF-ICE patient population
3. The potential long-term medical outcome effects of the additional ARTICE treatment compared to standard treatment alone.
4. The potential long-term health-related quality-of-life effects of ReActIF-ICE patient population
5. The potential long-term health-related quality-of-life effects of the additional ARTICE treatment compared to standard treatment alone.

In this long term follow up study, the enrolled subjects shall be followed up beyond 90 days for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal surrogate is willing and able to provide written informed consent and comply with all protocol requirements or the implementation of other established procedures according to the local regulations of the contributing center to include subjects who are unable to provide informed consent.
2. Subject was enrolled in the ReActIF-ICE study and successfully passed the Day 2 re-evaluation of that trial.

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All applicable subjects previously enrolled in the ReActIF-ICE study will be asked to participate in this long-term study, if they are fulfilling all inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Long term outcome after severe sepsis | 5 years
  Outcome evaluation parameters
  * Survival rates at 6 months,1,2,3,4,5 years
  * Serious Adverse Events rate during the 5 year follow up period

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Klinikum Magdeburg, Klinik für Intensiv- und Rettungsmedizin, Magdeburg
  - Universitätsmedizin Rostock, Abteilung KAI, Rostock

IPD SHARING:
Plan to Share IPD: No